CLINICAL TRIAL: NCT07120841
Title: Evaluation the Effect of "Nurse Telephone Follow-up" on Depression, Anxiety and Stress and Readmission of Cardiovascular Patients in Hospitalized Patients in Mazandaran Province
Brief Title: Nurse Telephone Follow-up for Cardiovascular Patients
Acronym: Nurse-TEL-CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hossein Mohsenipouya, Assistant professor of health education and promotion, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IR.MAZUMS.REC.1401.269; IR.MAZUMS.REC.1401.269 (Other: Mazandaran University of Medical Sciences, Ethics Committee)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Depression, Anxiety Disorders; Follow-up Study; Cardiovascular Diseases
Keywords: Cardiovascular patients; Depression, Anxiety, Stress; Telephone follow-up nursing
MeSH Terms: conditions — Depression; Anxiety Disorders; Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a parallel assignment to intervention and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients receive telephone follow-up education by nurse.
  Interventions: Behavioral: Telephone Education
- Control Group (Active Comparator): Patients receive usual care without follow-up education.
  Interventions: Behavioral: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Telephone Education — Participants in this group will receive telephone follow-up education by a nurse during the two weeks after discharge
  Arms: Intervention Group
Behavioral: Standard Care (in control arm) — Participants in this group will receive standard post-discharge care without any follow-up telephone education
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effect of follow-up telephone education provided by a nurse on the levels of anxiety, stress, and depression in patients hospitalized in the cardiac intensive care unit during the two weeks after discharge. Patients will be randomly assigned to either the intervention (education) group or the control group. Their levels of anxiety, stress, and depression will be measured before and after the intervention. The aim is to determine whether this educational intervention can improve the psychological well-being of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained from both the patient and their family.
2. Definite diagnosis of heart disease confirmed by a specialist physician.
3. No previous history of psychological problems, based on the patient's medical records.
4. No prior participation in similar educational programs.

Exclusion Criteria:

1. Non response to the nurse's follow-up calls.
2. Failure to complete the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — No restriction based on gender identity.
Enrollment: 60 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety, stress Score(DASS-21) | 2 weeks after discharge
  Changes in depression, anxiety, stress scores as measured by DASS-21

CONTACTS AND LOCATIONS:
Locations (1):
- Khatam Hospital, Behshahr, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study